CLINICAL TRIAL: NCT02472613
Title: Comparison of Acupuncture and Fluoxetine for of Ischemic Post-stroke Depression：A Multicentre Randomized Controlled Trial
Brief Title: Acupuncture for Ischemic Post-stroke Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Collaborators: State Administration of Traditional Chinese Medicine of the People's Republic of China (Other Government); Tianjin Academy of Tradional Chinese Medicine Afflicated Hospital (Unknown); Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Prof Zhang Chunhong, State Administration of Traditional Chinese Medicine of the People's Republic of China, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201407001-6B
Record Dates: First submitted 2015-06-08; First posted 2015-06-16 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Post-stroke Depression
Keywords: Post-Stroke Depression; Acupunture; Fluoxetine; RCT
MeSH Terms: interventions — Acupuncture Therapy; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- traditional acupuncture & placebo (Experimental): Apply traditional acupuncture to treat the ischemic post-stroke depression according to TCM theory.
  Interventions: Device: acupuncture; Drug: placebo
- sham-acupoint acupuncture & fluoxetine (Active Comparator): Fluoxetine was given at a dose of 20 mg/day. sham-acupoint will be penetrated for treat the ischemic post-stroke depression.
  Interventions: Device: sham-acupoint acupuncture; Drug: Fluoxetine

INTERVENTIONS:
Device: acupuncture — Patients will be treated at Renzhong（Du26）, Yintang（EX-HN3）、accupuncture Shangxing（DU23）penetrate to Baihui（DU20）,Sishencong（EX-HN1）; Neiguan（PC6）,Sibai（ST2）,Fengchi（GB20）and Sanyinjiao（SP6）in bilateral;Jianyu（LI15）,Quchi（LI11）,Shousanli（LI10）,Hegu（LI 4）, Fengshi (GB31),Xuehai（SP10） ,Zusanli（ST36）、Taichong（LR 3） of the hemiplegia side. There are another six groups of acupoints in bilateral. The acupuncturist will choose one group acupoints according to patients syndrome:Zhigou (SJ6),Qimen (LR14);Xingjian (LR2),Xiaxi(GB43);Fenglong (ST40),Lianquan(RN23);Tongli (HT5),Xinshu (BL15);Xinshu (BL15),Pishu(BL20);Shenshu (BL23),Taixi (KI3).
  The acupoints are inserted at the depth of 20-30mm except Renzhong（Du26）, Sibai（ST2）, Sishencong（EX-HN1）are inserted at the depth of 5-10mm. The needles will be left for 30 minutes and then removed. Acupuncture treatment will consist of three sessions per week for 12 consecutive weeks.
  Arms: traditional acupuncture & placebo
Drug: placebo — Placebo was given for 12 consecutive weeks.
  Arms: traditional acupuncture & placebo
Device: sham-acupoint acupuncture — Jianliao（SJ14）,Tianquan（PC2）,Xiabai (LU4),Xiaoluo (SJ12),Shouwuli (LI13),Sidu (SJ9),Huizong (SJ7),Wenliu (LI7),Zhouliao (LI12),Quze（PC3）,Kongzui（LI6）,Zhigou（SJ6）,Zhongzhu（SJ3）,Futu（ST32）,Jimen (SP11),Yinshi (ST33),Liangqiu（ST34）,Shangjuxu（ST37）,Xiajuxu（ST39）,Xiyangguan（GB33）,Ligou（LR5）,Pucan (BL61),Jinggu (BL64),Rangu (KI2),Ligou (LR5),Neiting （ST44） of the hemiplegia side.
  • The acupoints are inserted at the depth of 20-30mm,except Pucan (BL61),Jinggu (BL64),Rangu (KI2) ,Neiting （ST44）are inserted at the depth of 5-10mm. The needles will be left for 30 minutes and then removed. Acupuncture treatment will consist of three sessions per week for 12 consecutive weeks.
  Arms: sham-acupoint acupuncture & fluoxetine
Drug: Fluoxetine — Fluoxetine was given at a dose of 20 mg/day for12 consecutive weeks.
  Arms: sham-acupoint acupuncture & fluoxetine

SUMMARY:
This is a multicentre, single Blind ,randomized controlled clinical trial in ischemic post-stroke depression patients.The participants will be allocated randomly in either of the two groups: verum acupuncture plus placebo medication group or sham acupuncture plus true medication group. On the hypothesis that acupuncture intervention could produce the same therapeutic effects as antidepressants. The investigators also hypothesized that acupuncture would be associated with minimal side effects.

DETAILED DESCRIPTION:
Aim: To observe the curative effect of acupuncture in the treatment of Ischemic Post-Stroke Depression． Design: A multicentre,open-label randomized controlled trial will be performed in Tianjin and Beijing . Two hundred and eight participants with Ischemic Post-Stroke Depression patients were randomly divided into two groups which were both given basic treatment of stroke. The acupuncture group was given Tiaoshenkaiqiao acupuncture therapy and placebo，while the control group was treated with fluoxetine tablets and sham acupoint acupuncture treatment. Evaluated the clinical efficacy of the two groups with Hamilton Depression Scale(HAMD), Barthel Index (BI),Treatment Emergent Symptom Scale,(TESS ),Clinical Global Impression Scale(CGI) respectively before treatment, the second weekend of treatment ,the fourth weekend of treatment, the eighth weekend of treatment, the twelfth weekend of treatment. And observed the adverse reaction of the two groups.

Each participants will receive 36 sessions of acupuncture in 12 weeks, with a duration of 30 minutes in a session. After all the treatments were accomplished, there will be one follow-ups in the 24th week.

ELIGIBILITY:
Inclusion Criteria:

* in accordance with diagnosis of ischemic stroke in International Classification of Diseases-10 163, （ICD-10 163）;
* diagnosis of a major depressive episode according to the depression module of the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders-IV （DSM-IV）or Chinese Classification and Diagnostic Criteria of Mental Disorders-3(CCMD-3)
* age of a subject is between 40 and 80 years old, male or female;
* most recently experience an ischemic post-stroke depression and recent (<6 months);
* conscious, examination cooperation, without aphasia and severe cognitive impairment;
* capacity to provide written consent for both research assessment and treatment.

Exclusion Criteria:

* participation in any clinical trial within the previous or taking antidepressant treatment 2 weeks prior to baseline;
* presence of severe cognitive dysfunction, indicated the Mini-mental State Examination (MMSE) score of < 17
* presence of severe aphasia;
* had a history of psychiatric illness or depression
* impaired hepatic , renal function., hematological systems and so on;
* those who can not cooperate with treatment;
* pregnant women or women in lactation
* presence of another chronic disorder, including chronic alcoholism or durg abuse

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Depression Scale( HAMD-17) | 12 weeks
  Depression symptoms are primarily measured using the 17-item Hamilton Depression Scale (HAMD-17)
Barthel Index (BI) | 12 weeks
  physical outcomes will be measured using Barthel Index (BI)
Clinical Global Impression (CGI) | 12 weeks
  Clinical Global Impression (CGI) would also be measured by clinician

SECONDARY OUTCOMES:
Self-Rating Depression Scale(SDS) | 12 weeks
Treatment Emergent Symptom Scale,(TESS ) | 12 weeks
Stroke diagnosis and evaluation criteria of Traditional Chinese Medicine（TCM） | 12 weeks

OTHER OUTCOMES:
Ratio of NAA/Cr，Cho/Cr，mI/Cr by Magnetic Resoance Spectroscopy(MRS) | 12 weeks
  Compare the ratio of NAA/Cr，Cho/Cr，mI/Cr in brain bilateral dorsolateral prefrontal, anterior cingulate alter brain metabolism after treatment.
Determination of the content change of cytokines IL-1β, IL-6, TNF-α, BDNF in plasma | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - First Affiliated hospital of Tianjin University of TCM, Tianjin, Tianjin Municipality
  - Tianjin Academy of Tradional Chinese Medicine Afflicated Hospital, Tianjin, Tianjin Municipality
  - Beijing Hospital of Traditional Chinese Medicine, Beijing